CLINICAL TRIAL: NCT00005119
Title: Altered Calcium And Vitamin D Metabolism in PMDD
Brief Title: Altered Calcium and Vitamin D in PMDD or Severe PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Model: Parallel | Purpose: Diagnostic
Other Study IDs: STHYS-JACOBS (completed); DK57869-01
Record Dates: First submitted 2000-04-19; First posted 2000-04-20 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Dysphoric Disorder; Severe Premenstrual Syndrome; Calcium metabolism; Vitamin D; Bone Markers; Premenopausal; Menstrual Cycle
MeSH Terms: conditions — Premenstrual Syndrome; Premenstrual Dysphoric Disorder | interventions — Bone Remodeling

INTERVENTIONS:
Procedure: Measures of calcium and bone turnover

SUMMARY:
Osteoporosis has become one of the most widely recognized disorders of our times affecting an estimated 25 million women in this country. Recent evidence has suggested that premenstrual syndrome (PMS) is associated with a calcium deficiency state and bone loss. This may place premenopausal women at greater risk for osteoporosis. An entity such as PMS may be an important physiological marker of a calcium disturbance. The purpose of this investigation is to understand more completely the extent to which calcium balance is disturbed in severe PMS or Premenstrual Dysphoric Disorder (PMDD) by utilizing new tools to assess calcium and bone turnover. The long term objective is to elucidate the pathophysiology of PMDD or severe PMS as it relates to calcium hormones and bone markers. The experimental design involves the comparison between women witn severe PMS and asymptomatic controls.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of severe PMS for the PMS group
* No medical history of PMS for the control group
* Prospective 2 month documentation of moderate to severe symptoms for the PMS group
* Prospective 2 month documentation of absent symptoms for the control group
* General good health
* Regular menstrual cycles
* No history of metabolic bone disease

Exclusion Criteria:

* Amenorrhea
* Anorexia nervosa
* Malabsorption
* Inflammatory bowel disease
* Erosive gastrointestinal disease
* Gastrectomy
* Malignancy
* Multiple myeloma
* Primary hyperparathyroidism
* Use of suppressive doses of thyroxine
* Cushing's syndrome
* Use of glucocorticoids or anticonvulsants
* Use of diuretics
* Metabolic bone disease
* Pregnancy or perimenopause or menopause
* Mental retardation
* Menstrual irregularity
* Significant gynecologic abnormality
* Use of birth control pills

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2000-05; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Susan Thys-Jacobs, MD, Principal Investigator — St.Luke's-Roosevelt Hospital- Columbia Presbyterian Medical Center
Locations (1):
- St. Luke's-Roosevelt Hospital, New York, New York, United States

REFERENCES:
- [Background] Thys-Jacobs, Silverton M, Alvir JM et al. Reduced Bone Mass in women with Premenstrual Syndrome. J Women's Health 1995; 4:161.
- [Background] Thys-Jacobs S, Ceccarelli S, Bierman A, Weisman H, Cohen MA, Alvir J. Calcium supplementation in premenstrual syndrome: a randomized crossover trial. J Gen Intern Med. 1989 May-Jun;4(3):183-9. doi: 10.1007/BF02599520. PMID 2656936
- [Background] Thys-Jacobs S, Starkey P, Bernstein D, Tian J. Calcium carbonate and the premenstrual syndrome: effects on premenstrual and menstrual symptoms. Premenstrual Syndrome Study Group. Am J Obstet Gynecol. 1998 Aug;179(2):444-52. doi: 10.1016/s0002-9378(98)70377-1. PMID 9731851
- [Background] Thys-Jacobs S, Alvir MJ. Calcium-regulating hormones across the menstrual cycle: evidence of a secondary hyperparathyroidism in women with PMS. J Clin Endocrinol Metab. 1995 Jul;80(7):2227-32. doi: 10.1210/jcem.80.7.7608284.
- [Background] Lee SJ, Kanis JA. An association between osteoporosis and premenstrual symptoms and postmenopausal symptoms. Bone Miner. 1994 Feb;24(2):127-34. doi: 10.1016/s0169-6009(08)80150-x. PMID 8199532